CLINICAL TRIAL: NCT03085914
Title: A Phase 1/2, Open-Label, Safety, Tolerability, and Efficacy Study of Epacadostat in Combination With Pembrolizumab and Chemotherapy in Subjects With Advanced or Metastatic Solid Tumors (ECHO-207/KEYNOTE-723)
Brief Title: A Study of Epacadostat in Combination With Pembrolizumab and Chemotherapy in Participants With Advanced or Metastatic Solid Tumors (ECHO-207/KEYNOTE-723)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-207 / ECHO-207; 2016-004678-16 (EudraCT Number)
Record Dates: First submitted 2017-02-28; First posted 2017-03-21 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor
Keywords: solid tumors; colorectal cancer; pancreatic ductal adenocarcinoma; non-small cell lung cancer; PD-1; PD-L1; epacadostat; IDO inhibitor
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — epacadostat; pembrolizumab; Oxaliplatin; Leucovorin; Fluorouracil; Gemcitabine; 130-nm albumin-bound paclitaxel; Carboplatin; Paclitaxel; Pemetrexed; Cyclophosphamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Treatment Group A (Experimental): Epacadostat + pembrolizumab + mFOLFOX6 (oxaliplatin, leucovorin, 5-fluorouracil)
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- Treatment Group B (Experimental): Epacadostat + pembrolizumab + gemcitabine and nab-paclitaxel
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Gemcitabine; Drug: nab-Paclitaxel
- Treatment Group C (Experimental): Epacadostat + pembrolizumab + carboplatin and paclitaxel
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel
- Treatment Group D (Experimental): Epacadostat + pembrolizumab + pemetrexed and investigators choice of platinum agent
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Investigator's choice of platinum agent
- Treatment Group E (Experimental): Epacadostat + pembrolizumab + cyclophosphamide
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Cyclophosphamide
- Treatment Group F (Experimental): Epacadostat + pembrolizumab + gemcitabine and investigators choice of platinum agent
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Gemcitabine
- Treatment Group G (Experimental): Epacadostat + pembrolizumab + investigators choice of platinum agent and 5-fluorouracil
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-Fluorouracil; Drug: Investigator's choice of platinum agent

INTERVENTIONS:
Drug: Epacadostat — Epacadostat oral twice-daily continuous daily dosing at the protocol-defined dose.
  Other Names: INCB024360
Drug: Pembrolizumab — Pembrolizumab
Drug: Oxaliplatin — Oxaliplatin
  Arms: Treatment Group A
Drug: Leucovorin — Leucovorin
  Arms: Treatment Group A
Drug: 5-Fluorouracil — 5-Fluorouracil
  Arms: Treatment Group A
Drug: Gemcitabine — Gemcitabine
  Arms: Treatment Group B; Treatment Group F
Drug: nab-Paclitaxel — nab-Paclitaxel
  Arms: Treatment Group B
Drug: Carboplatin — Carboplatin
  Arms: Treatment Group C
Drug: Paclitaxel — Paclitaxel
  Arms: Treatment Group C
Drug: Pemetrexed — Pemetrexed
  Arms: Treatment Group D
Drug: Cyclophosphamide — Cyclophosphamide
  Arms: Treatment Group E
Drug: Carboplatin — Carboplatin
  Arms: Treatment Group D; Treatment Group G
Drug: Cisplatin — Cisplatin
  Arms: Treatment Group D; Treatment Group G
Drug: 5-Fluorouracil — 5-FU
  Arms: Treatment Group G
Drug: Investigator's choice of platinum agent — Investigator's choice of platinum agent: carboplatin or cisplatin
  Arms: Treatment Group D; Treatment Group G

SUMMARY:
This was an open-label, nonrandomized, Phase 1/2 study designed to determine the safety, tolerability, and efficacy of epacadostat when given in combination with pembrolizumab and 7 different chemotherapy regimens described as Treatment Groups A through G below (see Study Drug and Background Therapies, Dose, and Mode of Administration). Phase 1 consisted of a 3 + 3 + 3 design intended to determine the MTD or PAD of epacadostat when given in combination with pembrolizumab and chemotherapy; efficacy was also explored.

Phase 2 was designed to enroll efficacy expansion cohorts to further evaluate the safety, tolerability, and efficacy of epacadostat at the MTD or PAD (as selected in Phase 1) when given in combination with pembrolizumab and chemotherapy. Each efficacy expansion cohort was to enroll participants with 1 specific type of advanced or metastatic solid tumor. Additional cohorts (ie, the mandatory biopsy cohorts) were designed to evaluate changes in the tumor microenvironment in participants with any advanced or metastatic solid tumor who had progressed on previous therapy with a PD-1 or a PD-L1 inhibitor.

No participants were enrolled in any Phase 2 efficacy expansion cohort, or in any Phase 2 mandatory biopsy cohort receiving Treatment A, B, F, or G. Phase 2 mandatory biopsy cohort participants received Treatments C, D, or E (ie, were included in Treatment Groups C, D, or E). Participants were assigned to a treatment group based on the chemotherapy regimen most appropriate for their tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of selected advanced or metastatic solid tumors.
* Presence of measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the Protocol-defined range.
* Receipt of anticancer medications or investigational drugs within the Protocol-defined intervals before the first administration of study drug.
* Previous radiotherapy within 2 weeks of starting study therapy.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has not recovered to ≤ Grade 1 from toxic effects of previous therapy and/or complications from previous surgical intervention before starting study therapy.
* Receipt of a live vaccine within 30 days of planned start of study therapy.
* Active infection requiring systemic therapy.
* Subjects who have any active or inactive autoimmune disease or syndrome.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina Bio-Oncology Institute, PLLC, Huntersville, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Tennessee Oncology - Nashville; The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University; Henry Joyce Cancer Clinic, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Powderly JD, Klempner SJ, Naing A, Bendell J, Garrido-Laguna I, Catenacci DVT, Taylor MH, Lee JJ, Zheng F, Zhou F, Gong X, Gowda H, Beatty GL. Epacadostat Plus Pembrolizumab and Chemotherapy for Advanced Solid Tumors: Results from the Phase I/II ECHO-207/KEYNOTE-723 Study. Oncologist. 2022 Nov 3;27(11):905-e848. doi: 10.1093/oncolo/oyac174. PMID 36156099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 study sites in the US. Phases 1 and 2 each consisted of Treatment Groups A-G, and every patient in the same group in Phases 1 and 2 received the same dose of epacadostat (100 mg BID oral), pembrolizumab (200 mg IV), and the respective chemotherapy regimens. Data analysis and summarization were performed by treatment group, by combining data of the same group in Phases 1 and 2.
Pre-assignment Details: A total of 70 participants were enrolled in the study. Study enrollment was permanently discontinued on 25 Oct 2018 as a strategic decision. At the time of data cut-off date of 25 Jan 2019, 11 participants were ongoing on treatment. . Phase 2 consisted of efficacy expansion and Mandatory biopsy cohorts. Phase 2 Efficacy expansion cohorts did not open for enrollment. Phase 2/Mandatory biopsy cohorts opened for enrollment and only groups C, D and E enrolled participants prior to study termination
Groups:
- Group A: Epa + Pembrolizumab +mFOLFOX6: Epacadostat (Epa, 100 mg ) oral twice-daily (BID) continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg)administered intravenously (IV) in combination with mFOLFOX6 (oxaliplatin IV + leucovorin IV + 5-fluorouracil (5-FU) IV.
- Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with nab-paclitaxel IV and gemcitabine IV.
- Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) in combination with paclitaxel IV and carboplatin IV.
- Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with pemetrexed IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
- Group E: Epa + Pembrolizumab + Cyclophosphamide: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with cyclophosphamide PO.
- Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent: Epa (100mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with gemcitabine IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
- Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with 5-FU IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
Period: Overall Study
Arm/Group | Group A: Epa + Pembrolizumab +mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent
Started | 9 | 9 | 11 | 9 | 13 | 8 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 9 | 11 | 9 | 13 | 8 | 11
Not completed — Death | 6 | 6 | 4 | 1 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Reason was not specified, | 2 | 2 | 2 | 3 | 3 | 3 | 6
Not completed — Progressive Disease | 0 | 0 | 2 | 2 | 1 | 1 | 1
Not completed — Study Terminated by the Sponsor | 0 | 0 | 0 | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants enrolled in the study who received at least 1 dose of epacadostat, pembrolizumab, or an applicable chemotherapy regimen.
Groups:
- Group A: Epa + Pembrolizumab + mFOLFOX6: Epacadostat (Epa) oral twice-daily (BID) continuous daily dosing at the protocol-defined dose in combination with pembrolizumab administered intravenously (IV) in combination with mFOLFOX6 (oxaliplatin IV + leucovorin IV + 5-fluorouracil (5-FU) IV.
- Group E: Epa + Pembrolizumab + Cyclophosphamide: Epa (100 mg)oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with cyclophosphamide PO.
- Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent: Epa (100 mg) oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with gemcitabine IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
- Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent: Epa (100 mg) oral BID continuousdaily dosing at the protocol-defined dose in combination with pembrolizumab (200 mg) IV in combination with 5-FU IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
- Total: Total of all reporting groups
Arm/Group | Group A: Epa + Pembrolizumab + mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent | Total
Number analyzed (Participants) | 9 | 9 | 11 | 9 | 13 | 8 | 11 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (8.03) | 46.0 (14.98) | 63.7 (12.11) | 58.2 (12.96) | 62.0 (10.21) | 60.3 (12.01) | 59.4 (12.24) | 58.3 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 4 | 10 | 5 | 4 | 36
  Male | 6 | 5 | 5 | 5 | 3 | 3 | 7 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 7 | 7 | 9 | 8 | 10 | 6 | 8 | 55
  Race: Black/African-American | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 6
  Race: Asian | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
  Race: Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race: Other | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Ethnicity: Not Hispanic or Latino | 9 | 9 | 11 | 7 | 13 | 8 | 10 | 67
  Ethnicity: Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Ethnicity: Unknown | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phases 1 & 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of epacadostat, pembrolizumab, or chemotherapy. Serious adverse event is defined as an event that meets 1 of the following criteria: is fatal or life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability, incapacity, or a substantial disruption of a person's ability to conduct normal life functions, constitutes a congenital anomaly or birth defect,is a medically important event that may jeopardize the participant or may require medical or surgical intervention to prevent 1 of the outcomes listed above.
Time Frame: Up to 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent: Epa oral BID continuous daily dosing at the protocol-defined dose in combination with pembrolizumab IV in combination with gemcitabine IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
- Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent: Epa oral BID continuousdaily dosing at the protocol-defined dose in combination with pembrolizumab IV in combination with 5-FU IV and Investigator's choice of platinum agent: carboplatin IV or cisplatin IV.
Arm/Group | Group A: Epa + Pembrolizumab + mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent
Number analyzed (Participants) | 9 | 9 | 11 | 9 | 13 | 8 | 11
Participants
  TEAE | 9 | 9 | 11 | 9 | 13 | 8 | 11
  Serious TEAE | 5 | 5 | 3 | 6 | 4 | 6 | 5

2. Primary Outcome: Phases 1 and 2: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any of the protocol-specified toxicities occurring up to and including Day 28 for the cohorts where mFOLFOX6 and nab-paclitaxel/gemcitabine are administered and Day 21 for all other chemotherapy regimens in Phase 1, except those with a clear alternative explanation (eg, disease progression) or transient (≤ 72 hours) abnormal laboratory values without associated clinically significant signs or symptoms based on investigator determination.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Epa + Pembrolizumab + mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent
Number analyzed (Participants) | 9 | 9 | 11 | 9 | 13 | 8 | 11
Participants | 2 | 0 | 0 | 0 | 0 | 3 | 0

3. Primary Outcome: Phases 1 and 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Up to Week 18
Population: The full analysis set included all participants enrolled in the study who received at least 1 dose of epacadostat and have at least 1 postbaseline assessment or who discontinued epacadostat.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Epa + Pembrolizumab + mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent
Number analyzed (Participants) | 9 | 9 | 11 | 9 | 13 | 8 | 11
Participants
  Complete Response | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Partial Response | 5 | 2 | 3 | 2 | 3 | 1 | 5

ADVERSE EVENTS:
Time Frame: Up to 21 months
Description: The safety population included all participants enrolled in the study who received at least 1 dose of epacadostat, pembrolizumab, or an applicable chemotherapy regimen.
Groups:
- Total: Total
Arm/Group | Group A: Epa + Pembrolizumab + mFOLFOX6 | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent | Group E: Epa + Pembrolizumab + Cyclophosphamide | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent | Total
All-Cause Mortality (participants affected / at risk) | 6/9 | 6/9 | 4/11 | 1/9 | 6/13 | 2/8 | 3/11 | 28/70
Serious Adverse Events (participants affected / at risk) | 5/9 | 5/9 | 5/11 | 3/9 | 6/13 | 4/8 | 6/11 | 34/70
Other Adverse Events (participants affected / at risk) | 9/9 | 8/9 | 11/11 | 9/9 | 13/13 | 8/8 | 10/11 | 68/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Epa + Pembrolizumab + mFOLFOX6 (N=9) | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine (N=9) | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin (N=11) | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent (N=9) | Group E: Epa + Pembrolizumab + Cyclophosphamide (N=13) | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent (N=8) | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent (N=11) | Total (N=70)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ammonia increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Disease progression (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pure white cell aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Epa + Pembrolizumab + mFOLFOX6 (N=9) | Group B: Epa + Pembrolizumab + Nab-Paclitaxel and Gemcitabine (N=9) | Group C: Epa + Pembrolizumab + Paclitaxel and Carboplatin (N=11) | Group D: Epa + Pembrolizumab + Pemetrexed and Platinum Agent (N=9) | Group E: Epa + Pembrolizumab + Cyclophosphamide (N=13) | Group F: Epa + Pembrolizumab + Gemcitabine and Platinum Agent (N=8) | Group G: Epa + Pembrolizumab + 5-FU and Platinum Agent (N=11) | Total (N=70)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (16)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 8 (9)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 16 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (9)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (6) | 4 (5) | 3 (4) | 6 (9) | 4 (4) | 3 (3) | 27 (33)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorectal swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 7 (8)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (4) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 14 (16)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Bacteroides bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 13 (13)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (8)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 10 (11)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 9 (10)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 13 (15)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 12 (13)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 13 (15)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 5 (6) | 6 (6) | 4 (4) | 4 (5) | 0 (0) | 4 (5) | 26 (32)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 5 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (9) | 5 (7) | 6 (7) | 7 (7) | 6 (6) | 4 (4) | 4 (4) | 39 (44)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Head titubation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 9 (9)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 2 (3) | 0 (0) | 1 (1) | 10 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 10 (10)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 3 (3) | 2 (2) | 1 (1) | 4 (8) | 1 (1) | 13 (20)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 11 (12)
Malaise (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (5) | 8 (13) | 7 (7) | 4 (5) | 4 (4) | 7 (7) | 37 (44)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 7 (8) | 3 (4) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 19 (21)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 5 (13) | 5 (5) | 2 (2) | 2 (5) | 5 (9) | 3 (3) | 24 (44)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1) | 3 (6) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 8 (13)
Neutrophil toxic granulation present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (4)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (8)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (9)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 10 (11)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
Pyuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 14 (17)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal salt-wasting syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shift to the left (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site irritation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 5 (7) | 16 (20)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (16) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 2 (3) | 15 (26)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 5 (6)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 6 (6)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 3 (4) | 3 (3) | 3 (3) | 20 (21)
Vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
White blood cell count decreased (Investigations) | 1 (2) | 1 (1) | 3 (7) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 9 (16)

LIMITATIONS AND CAVEATS:
Enrollment in this study was permanently discontinued on 25 Oct 2018 due to a strategic decision and not based on safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03085914/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03085914/SAP_001.pdf